CLINICAL TRIAL: NCT03464565
Title: COMPLETE: International Acute Ischemic Stroke Registry With the Penumbra System Aspiration Including the 3D Revascularization Device
Status: Completed | Type: Observational
Sponsor: Penumbra Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 12965
Record Dates: First submitted 2018-03-07; First posted 2018-03-14 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Stroke, Ischemic
Keywords: Large Vessel Occlusion; Acute Ischemic Stroke; Mechanical Thrombectomy; Penumbra System; 3D Revascularization
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patients with acute ischemic stroke secondary to LVO
  Interventions: Device: Penumbra System

INTERVENTIONS:
Device: Penumbra System — Penumbra System

SUMMARY:
The purpose of this registry is to collect performance and safety data on the Penumbra System including the 3D Revascularization Device in a real world patient population with acute ischemic stroke (AIS) secondary to intracranial large vessel occlusion (LVO).

DETAILED DESCRIPTION:
Registry Objective: The primary objective of this registry is to collect real-world performance and safety data on Penumbra System including the 3D Revascularization Device in a patient population with acute ischemic stroke (AIS) secondary to intracranial large vessel occlusion (LVO).

Registry Design: This will be a prospective, single-arm, multi-center observational registry and will include patients that present with either anterior or posterior LVO who are eligible for mechanical thrombectomy using the Penumbra System.

Registry Duration: Subjects will be in the registry for approximately 90 days from enrollment to last follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥ 18
* Pre-stroke mRS 0-1
* Patient experiencing acute ischemic stroke secondary to intracranial large vessel occlusion who are eligible for mechanical thrombectomy using the Penumbra System
* Planned frontline treatment with Penumbra System
* Signed informed consent per Institution Review Board/Ethics Committee

Exclusion Criteria:

* Any comorbid disease or condition expected to compromise survival or ability to complete follow-up assessments through 90 days.
* Currently participating in an investigational (drug, device, etc) clinical trial that will confound study endpoints. Patients in observational, natural history, and/or epidemiological studies not involving intervention are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients experiencing acute ischemic stroke secondary to intracranial large vessel occlusion who are eligible for mechanical thrombectomy using the Penumbra System
Sampling Method: Non-Probability Sample
Enrollment: 650 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
mTICI Score | Post Procedure
  Angiographic revascularization of the occluded target vessel at immediate post-procedure as defined by a modified treatment in cerebral infarction (mTICI) score 2b or higher.
  mTICI scale ranges 0 to 3 higher values represent better outcomes.
Functional Subject Outcome | 90 days post
  Functional subject outcome at 90 days post-procedure as defined by a modified Rankin Scale (mRS) 0-2.
  mRS scale ranges 0 to 6 higher values represent a worse outcome.
All-cause mortality at 90 days | 90 days
  All-cause mortality at 90 days

SECONDARY OUTCOMES:
Incidence of device and procedure related Serious Adverse Events (SAEs) | Within 24 hours of procedure
Occurrence of embolization in previously uninvolved (or new) territories (ENT) | During Procedure
  Occurrence of embolization in previously uninvolved (or new) territories (ENT) as seen on the final control angiogram at the end of procedure
Occurrence of symptomatic intracranial hemorrhages (sICH) | 24 Hours Post Procedure
Time to Revascularization | During Procedure
Length of hospital stay | Through discharge, up to study completion at approximately 90 days
Discharge Facility | Through discharge, up to study completion at approximately 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Osama O Zaidat, MD, Principal Investigator — Mercy St. Vincent Medical Center; Johanna Fifi, MD, Principal Investigator — Mount Sinai Health System; Ameer E. Hassan, MD, Principal Investigator — McAllen Medical Center
Locations (42):
- United States (29):
  - Banner Desert Medical Center, Mesa, Arizona
  - Eden Medical Center, Castro Valley, California
  - St. Jude Medical Center, Fullerton, California
  - Cedar Sinai Medical Center, Los Angeles, California
  - Mercy San Juan Medical Center, Sacramento, California
  - Los Robles Hospital, Thousand Oaks, California
  - RIA, Englewood, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Jackson Memorial Hospital, Miami, Florida
  - Naples Community Hospital, Naples, Florida
  - AdventHealth Orlando, Orlando, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Oschner Medical Center, New Orleans, Louisiana
  - Brigham & Women's Hospital, Boston, Massachusetts
  - SSM St. Clare Healthcare, St Louis, Missouri
  - The Valley Hospital, Ridgewood, New Jersey
  - Northwell Health, Manhasset, New York
  - Mount Sinai New York, New York, New York
  - NYU Langone Hospital-Brooklyn, New York, New York
  - Mercy St. Vincent Medical Center, Toledo, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Palmetto Health Richland Hospital, Columbia, South Carolina
  - Erlanger Health System, Chattanooga, Tennessee
  - Fort Sanders Regional Medical Center, Knoxville, Tennessee
  - Methodist University Hospital, Memphis, Tennessee
  - Valley Baptist Medical Center, Harlingen, Texas
  - Houston Methodist Hospital, Houston, Texas
  - McAllen Medical Center, McAllen, Texas
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
- France (2):
  - CHU de Bordeaux - Hôpital Pellegrin, Bordeaux
  - Foundation Ophthalmic Adolphe De Rothschild, Paris
- Germany (5):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Schleswig-Holstein Campus Lübeck, Lübeck
  - Universitätsklinikum Magdeburg A. ö. R., Magdeburg
- Samodzielny Publiczny Szpital Kliniczny, Lublin, Poland
- Russia (3):
  - Davidovsky Moscow City Hospital №23, Moscow
  - City Clinical Hospital No. 1, Moscow
  - Multidisciplinary City Hospital №2, Saint Petersburg
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia

REFERENCES:
- [Derived] Hassan AE, Fifi JT, Zaidat OO. Aspiration thrombectomy with the Penumbra System for patients with stroke and late onset to treatment: a subset analysis of the COMPLETE registry. Front Neurol. 2023 Sep 14;14:1239640. doi: 10.3389/fneur.2023.1239640. eCollection 2023. PMID 37794880
- [Derived] Hassan AE, Zaidat OO, Nanda A, Atchie B, Woodward K, Doerfler A, Tomasello A, Fifi JT. Impact of interhospital transfer vs. direct admission on acute ischemic stroke patients: A subset analysis of the COMPLETE registry. Front Neurol. 2022 Aug 9;13:896165. doi: 10.3389/fneur.2022.896165. eCollection 2022. PMID 36016541
- [Derived] Zaidat OO, Fifi JT, Nanda A, Atchie B, Woodward K, Doerfler A, Tomasello A, Tekle W, Singh IP, Matouk C, Thalwitzer J, Jargiello T, Skrypnik D, Beuing O, Berge J, Katz JM, Biondi A, Bonovich D, Sheth SA, Yoo AJ, Hassan AE; COMPLETE Registry Investigators. Endovascular Treatment of Acute Ischemic Stroke With the Penumbra System in Routine Practice: COMPLETE Registry Results. Stroke. 2022 Mar;53(3):769-778. doi: 10.1161/STROKEAHA.121.034268. Epub 2021 Sep 22. PMID 34547927